# Official Project Title:

Developing Inclusive Youth: Promoting Intergroup Friendships and Inclusive Classrooms in Childhood

NCT: Not Yet Assigned

Date of Upload: October 14, 2022

UMD IRB Approval Effective August 31, 2022

### **University of Maryland College Park**


| Initials: | Date: |
|-----------|-------|



Department of Human Development and Quantitative Methodology 3943 Campus Drive, Suite 3304 College Park, MD 20742-1131 Melanie Killen, Ph.D. Office: 301.405.3176 Email: mkillen@umd.edu

#### Dear Parents or Guardians:

We invite your child to participate in a project conducted by the University of Maryland Social and Moral Development called *Developing Inclusive Youth*. The goal of this project is to evaluate a program designed to increase friendships and school belonging as well as facilitate positive discussions regarding diversity and inclusion in peer contexts. We have successfully implemented the program in 24 classrooms in MCPS. We would like to ask permission to include your son or daughter for this project.

Specifically, student participation in the program involves viewing animated, voice-over peer scenarios in a web-based curriculum tool. Students decide who to include when the characters are discussing an activity together such as playing a game at recess, doing a school project, watching a movie at home, or playing a game at the park. The situations are drawn from every-day encounters. Children decide how each character feels and the reasons for their decisions. There are two different classroom groups. For half of the classrooms participating students will take a survey twice, and for the other half students will take the survey plus use the web-based tool and participate in a teacher-led classroom discussion.

All children will be asked to complete a survey on their thoughts about topics of friendship, attitudes towards different groups, and general feelings of school belongingness, once at the beginning and once at the end of the study. This survey will take approximately 25 minutes for children to complete and is composed of questions interspersed with pictures. Trained research assistants from the University of Maryland will be present to answer any questions or concerns from children during survey administration.

Participation is strictly voluntary. All information is confidential. Please look over the description below. If you are willing to have your child participate in the project, please fill out the information in the survey.

The information from our past research and our work with children and schools has helped teachers, policy makers, counselors and school administrators design curriculum and interventions to promote mutual respect among children and positive social environments for all children. This current research project has been approved by the Institutional Review Board at the University of Maryland. We thank you, in advance, for reading this letter, and for your willingness to allow your daughter/son to participate.

Sincerely,

Melanie Killen, Ph.D.

Professor of Human Development and Quantitative Methodology

## **University of Maryland College Park**


| Project Title | Dramatina Dagitiya Eriandahina in Vayth | | |
|---|---|---|---|
| Project fille | Promoting Positive Friendships in Youth This research is being conducted by Dr. Melanie Killen at the University of Maryland, College Park. We are inviting | | |
| Purpose of the | your child to participate in an evaluation of a program designed to facilitate productive discussions regarding diversity | | |
| Study | and inclusion in peer contexts. | esigned to identitute productive discussi | ons regarding diversity |
| | Your child will be given a survey that will take approximately curriculum. Trained research assistants from the University of | | |
| | randomly assigned to one of two options: 1) Survey-only, or 2) Survey plus program and classroom discussion. All participants will fill out | | |
| Procedures | a short 25-minute study survey about peer relationships and school belonging, once at the beginning and once at the end of the project. For the program option, children will view 15-minute scenarios drawn from every-day school and home peer encounters. Children will be | | |
| | introduced to characters in the story and will be prompted to re- | spond to several questions and make predict | ions about what the characters |
| | should do. Following the scenario, children will engage in a she learned. | ort teacher-facilitated classroom discussions | about the story and what they |
| | There are no reasonably foreseeable risks to individuals | who participate in this study. All respo | nses will be stored in locked |
| Potential Risks | cabinets and on secure, password protected servers provided by the University of Maryland. In the unlikely event of a | | |
| & Discomforts | breach of confidentiality, there remains a minor risk that<br>their participant ID numbers. UMD generated IDs will be | | |
| | confidentiality. | is assigned to each emid participating in | the program to protect |
| Potential | There are no immediate benefits from participation in th | | |
| Benefits | workers will be able to learn from this research and use<br>Your child's name will not be attached to their response on the | | |
| | for clarity and analyses of children's exchanges. No identifiable | | |
| | discussions. Recordings will be de-identified, and after five ye<br>number. A description of this clinical trial will be available on | | |
| Confidentiality | not include information that can identify you. At most, the Web | site will include a summary of the results. | You can search the web site at |
| | any time. We will not share your child's answers with anyone,<br>this research project, your child's identity will be protected. All | | |
| | servers provided by the University of Maryland. Your child's in | nformation may be shared with representative | es of the University of |
| | Maryland, College Park or governmental authorities if your child or someone else is in danger or if we are required to do so by law. Your child's participation is completely voluntary. Your child can ask any questions at any time. Your child may decide to | | |
| Dialet te | | | |
| Right to Withdraw & | stop participating at any time and will not be penalized or lose any benefits. Participation is not a school or class requirement. If you decide to stop taking part in the study, if you have questions, concerns, or complaints, or if you need to | | |
| Questions | report an injury related to the research, please contact th | | |
| | Development & Quantitative Methodology, 3942 Car 301-405-3176. Email: <a href="mailto:mkillen@umd.edu">mkillen@umd.edu</a> | npus Dr., Suite 3504 College Park, M | 1D 20/42-1131. Telephone: |
| | If you have questions about your rights as a research par | | |
| Participant | University of Maryland College Park Institutional Revie | | |
| Rights | E-mail: irb@umd.edu; Telephone: 301-405-0678. This is Maryland, College Park IRB procedures for research inv | | o the University of |
| | Your signature indicates that you are at least 18 years of | age; you have read this consent form o | |
| Statement of<br>Consent | your questions have been answered to your satisfaction a research study. You will receive a copy of this signed co | | |
| Oonsent | sign your name below. Children: you will be asked if yo | | |
| | 1. Child's Name | 2. Child's birthday | 3. Today's Date |
| | | / / | 1 1 |
| | 4. Parent/Guardian Name | 5. Parent/Guardiar | n Signature |
| | 6. Child's Grade | 7. Child's Classroo | om Teacher |
| | The following questions are optional and are used to ensure to | hat we have a representative sample of parti | cipants. |
| 8. Child Gender: Girl: Boy: Other: | | | |
| 9. Language(s) Spoken at Home (check all that apply): | | | |
| English: Spanish: Other(s) (please write in): | | | |
| 10. Child Race/Ethnicity (check all that apply) | | | |
| Black/African-American: White/European-American: Latino/Hispanic: | | | |
| Asian-American/Pacific Islander: Native American: Multiracial/Multiethnic: Other: | | | |

## **University of Maryland College Park**


| 11. Please mark each parent or guardian's highest level of education: | | | | |
|---|---|---|---|---|
| Parent 1: Mother: | Father: | Other: | _ | |
| Parent 1's highest level of education: Didn't graduate high school: High school graduate/GED: | | | | |
| Some college: Bachelor's Degree: Graduate Degree: | | | | |
| Parent 2: Mother: | Father: | Other: | _ | |
| Parent 2's highest level of education: Didn't graduate high school: High school graduate/GED: | | | | |
| Some college: | Bachelor's Degre | e: | Graduate Degre | e: |